CLINICAL TRIAL: NCT00850382
Title: Open-Label, Multicenter Phase Ib/IIa Study For the Evaluation of Dasatinib (Sprycel™) Following Induction and Consolida-tion Therapy as Well as in Maintenance Therapy in Patients With Newly Diagnosed Core Binding Factor (CBF) Acute Myeloid Leukemia (AML)
Brief Title: Dasatinib (Sprycel™) in Patients With Newly Diagnosed Core Binding Factor (CBF) Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 11-08
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: CBF AML; Dasatinib; Core Binding Factor (CBF)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dasatinib; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental): Induction cycle(s):
  Patients will receive in cycle 1 induction therapy with daunorubicin 60 mg/m2/day administered on days 1 through 3 and cytarabine 200 mg/m2/day administered by continuous IV infusion daily for 7 days (days 1 through 7). Patients will receive dasatinib 100 mg QD on days 8-21. Patients not achieving CR or CRi at the end of cycle 1 will be evaluable to receive a second induction cycle identical in schedule and dosage to the first induction cycle.
  Consolidation Cycles 1, 2, 3, 4:
  Patients achieving CR or CRi at the end of cycle 1 will receive consolidation therapy for 4 cy-cles. Consolidation therapy consists of high-dose cytarabine 3 g/m2 (>60 years: 1 g/m2) q12h, d 1, 3, 5, administered intravenously over three hours. Patients will receive dasatinib 100 mg QD on days 6-28.
  Maintenance therapy:
  Patients completing consolidation therapy will continue to receive single agent dasatinib 100 mg QD for one year (or until relapse).
  Interventions: Drug: Dasatinib; Drug: daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Dasatinib — Induction cycle(s):
  Dasatinib 100 mg QD on days 8-21.
  Consolidation Cycles 1, 2, 3, 4:
  Patients will receive dasatinib 100 mg QD on days 6-28.
  Maintenance therapy:
  Patients completing consolidation therapy will continue to receive single agent dasatinib 100 mg QD for one year (or until relapse).
Drug: daunorubicin — Induction cycle(s):
  Daunorubicin 60 mg/m2/day administered on days 1 through 3
Drug: Cytarabine — Induction cycle(s):
  Cytarabine 200 mg/m2/day administered by continuous IV infusion daily for 7 days (days 1 through 7).
  Consolidation cycles 1, 2, 3, 4:
  Consolidation therapy consists of high-dose cytarabine 3 g/m2 (>60 years: 1 g/m2) q12h, d 1, 3, 5, administered intravenously over three hours.

SUMMARY:
This is a Phase Ib/IIa open-labeled multi-center trial evaluating the feasibility of dasatinib given after standard induction therapy with daunorubicin (DNR) and cytarabine (ARA-C), after consolidation therapy with high-dose cytarabine (HDAC), and as single agent in a one-year maintenance therapy in patients with newly diagnosed CBF AML.

82 patients with newly diagnosed CBF AML will be enrolled at AMLSG study centers.

All AML patients will be assessed for the CBF fusion genes via the central laboratory of the AMLSG within 48 hours of diagnosis of AML, and only patients with CBF AML will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Core binding factor (CBF) AML with molecular diagnosis of RUNX1-RUNX1T1 fusion transcript resulting from t(8;21)(q22;q22) (or a variant form) or of CBFB-MYH11 fusion transcript resulting from inv(16)(p13.1q22)/t(16;16)(p13.1;q22) as assessed in one of the central AMLSG reference laboratories.
* Age ≥ 18; there is no upper age limit.
* No prior chemotherapy for leukemia except hydroxyurea for up to 5 days during the diag-nostic screening phase.
* Non-pregnant and non-nursing. Due to the unknown teratogenic potential of dasatinib in humans, pregnant or nursing patients may not be enrolled. Women of childbearing poten-tial (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration. Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control - one highly effective method (e.g., IUD, hormonal, tubal ligation, or partner's vasectomy), and one additional effective method (e.g., latex condom, diaphragm, or cervical cap) - AT THE SAME TIME, at least four weeks before she begins dasatinib therapy. "Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months.
* Men must agree not to father a child and must use a latex condom during any sexual con-tact with women of childbearing potential while taking dasatinib and for 4 weeks after therapy is stopped, even if they have undergone a successful vasectomy.
* Signed written informed consent

Exclusion Criteria:

* Performance status WHO >2
* Pulmonary edema and/or pleural/pericardial effusion within 14 days of Day 1. If edema/effusion resolves to CTC Grade ≤ 1, patients can be treated with dasatinib.
* Patients with ejection fraction < 50% by echocardiography within 14 days of day 1
* Organ insufficiency (creatinine >1.5x upper normal serum level; bilirubin, AST or AP >2.5x upper normal serum level; heart failure NYHA III/IV; severe obstructive or restrictive ventilation disorder)
* Uncontrolled infection
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* Known positive for HIV
* Bleeding disorder independent of leukemia
* No consent for registration, storage and processing of the individual disease-characteristics and course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Feasibility as combined endpoint: Rate of ED/HD Rate of pleural/pericardial effusion grade 3/4 Rate of liver toxicity grade 3/4 that does not improve to <= grade 2 within 14 days after discontinuing responsible medication Rate of refractory disease | after 4 weeks

SECONDARY OUTCOMES:
Cumulative incidence of relapse (CIR) and death (CID) | After follow-up period of two years
Overall survival (os) | After follow-up period of two years

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Doehner, MD, Principal Investigator — University Hospital of Ulm
Locations (50):
- Austria (5):
  - Universitätsklinikum Innsbruck, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Elisabethinen Krankenhaus, Linz
  - Landeskliniken Salzburg, Salzburg
  - Hanuschkrankenhaus Wien, Vienna
- Germany (45):
  - Ubbo-Emmius Klinik Aurich, Aurich
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Duesseldorf, Düsseldorf
  - Kliniken Essen-Sued, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Städtische Kliniken Frankfurt Höchst, Frankfurt-Höchst
  - Medizinische Universitätsklinik, Freiburg im Breisgau
  - Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Klinik der Justus Liebig Universität, Giessen
  - Wilhelm- Anton- Hospital gGmbH, Goch
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikum Hanau gGmbH, Hanau
  - Klinikum Hannover Siloah, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitätsklinikum des Saarlandes, Homburg Saar
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Staedtisches Krankenhaus Kiel GmbH, Kiel
  - Caritas Krankenhaus Lebach, Lebach
  - Klinikum Lippe-Lemgo, Lemgo
  - Klinikum Luedenscheid, Lüdenscheid
  - Univ-Klinikum der Otto- von Guericke- Universität, Magdeburg
  - Universitätsklinikum der Johannes Gutenberguniversität Mainz, Mainz
  - Johannes Wesling Klinikum, Minden
  - Klinikum rechts der Isar der TU Muenchen, München
  - Klinikum Oldenburg, Oldenburg
  - Klinikum Passau, Passau
  - Elisabeth Krankenhaus, Recklinghausen
  - Krankenhaus der Barmherzigen Brueder, Regensburg
  - Caritas-Klinik St. Theresia, Saarbrücken
  - Klinikum Sindelfingen-Böblingen, Sindelfingen
  - Klinikum Stuttgart, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Medizinische Universitätsklinik Tuebingen, Tübingen
  - Universitätsklinik Ulm, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Helios Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Paschka P, Schlenk RF, Weber D, Benner A, Bullinger L, Heuser M, Gaidzik VI, Thol F, Agrawal M, Teleanu V, Lubbert M, Fiedler W, Radsak M, Krauter J, Horst HA, Greil R, Mayer K, Kundgen A, Martens U, Heil G, Salih HR, Hertenstein B, Schwanen C, Wulf G, Lange E, Pfreundschuh M, Ringhoffer M, Girschikofsky M, Heinicke T, Kraemer D, Gohring G, Ganser A, Dohner K, Dohner H. Adding dasatinib to intensive treatment in core-binding factor acute myeloid leukemia-results of the AMLSG 11-08 trial. Leukemia. 2018 Jul;32(7):1621-1630. doi: 10.1038/s41375-018-0129-6. Epub 2018 Apr 17. PMID 29720733